CLINICAL TRIAL: NCT06218875
Title: Assessment of Long Term, Endovascular AAA Intervention Using the GORE® EXCLUDER® Conformable AAA Endoprosthesis or Iliac Branch Endoprosthesis
Brief Title: Endovascular AAA Intervention Using the GORE® EXCLUDER® Conformable AAA Endoprosthesis or Iliac Branch Endoprosthesis
Status: Recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: TGR 23-02AA
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: AAA - Abdominal Aortic Aneurysm
Keywords: Aneurysm; Aneurysm Repair; Endovascular; EVAR; Endoprosthesis; Aortic; Aortic Repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- GORE® EXCLUDER® Conformable AAA Endoprosthesis (EXCC Device): Patients treated with the EXCC Device
- GORE® EXCLUDER® Iliac Branch Endoprosthesis (IBE Device): Patients treated with the IBE Device

SUMMARY:
A prospective, observational post-market registry collecting outcomes through a 10-year post procedure follow-up for patients treated with the GORE® EXCLUDER® Conformable AAA Endoprosthesis (EXCC Device) or the GORE® EXCLUDER® Iliac Branch Endoprosthesis (IBE Device) as a part of routine clinical practice.

DETAILED DESCRIPTION:
The purpose of the Gore Together Aortic Registry is to collect real-world data (RWD) for Gore aortic endovascular devices. Due to the nature of the program, patient selection, diagnostic imaging, and treatment interventions will be determined by physicians based on standard clinical practice. Therefore, the Sponsor will not be outlining requirements that would influence healthcare decisions.

Participants will be asked to return for regular scheduled visits as requested by their surgeon. Patients will report any issues they may have regarding the device or surgery to their surgeon/doctor.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative (LAR) provides written authorization and/or consent per institution and geographical requirements
2. Patient has been or is intended to be treated with an eligible registry device
3. Patient is age ≥ 18 years at time of informed consent signature.

Exclusion Criteria:

1. Patient who is, at the time of consent, unlikely to be available for standard of care (SOC) follow-up visits as defined by the site's guidelines and procedures.
2. Patient with exclusion criteria required by local law.
3. Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study within 12 months of Together Registry enrollment. Subjects cannot be enrolled in another Together Registry module protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry participants are derived from patients presenting with vascular disease that may benefit from the placement of an endovascular stent graft. The target registry population is patients who are treated with either EXCC or IBE Device at participating sites. This includes initial procedures and reinterventions (regardless of original intervention). Only patients who meet all the inclusion and none of the exclusion criteria will be included in the registry.
  The registry has been designed with broad eligibility criteria to optimize the visibility of overall registry device use. An integral requirement to the target subject population is that the decision to use a GORE® EXCLUDER® product has been made prior to considering the patient for possible registry participation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2042-09-30 (Estimated); Study Completion 2042-09-30 (Estimated)

PRIMARY OUTCOMES:
Deployment Technical Success | Time of Surgery
  Successful access, delivery, and accurate deployment of the device to the intended location, and retrieval of the delivery system.
Lesion-related Mortality | Day 30 through Year 10
  Death related to the index endovascular procedure, secondary procedure associated with the index lesion or the registry device, or any death where the treated disease / index lesion or registry device caused or significantly contributed to the death
Lesion Rupture | Time of Surgery through Year 10
  Rupture in the treated segment of the vessel (e.g., aorta or branch) verified with direct observation or Computed Tomographic Angiography (CTA) scan
Lesion Enlargement | Time of Surgery through Year 10
  An increase in maximum vessel (e.g., aorta or treated branch) diameter of > 5 mm in the region encompassed by the initial lesion as compared to baseline using orthogonal (i.e., perpendicular to the centerline) measurements on CTA scans
Endoleaks | Time of Surgery through Year 10
  Perfusion of a treated lesion identified through imaging analysis
Device Migration | Time of Surgery through Year 10
  Longitudinal movement of all or part of the device for a distance ≥ 10 mm, as confirmed by CTA scan, relative to anatomical landmarks and device positioning at the first post-operative CTA scan.
Loss of aortic / branch patency | Time of Surgery through Year 10
  No flow or contrast detected through the implanted aortic and/or branch component (for branched devices) confirmed with imaging and/or direct observation.
New onset renal failure | Time of Surgery through Day 30
  New onset sustained renal failure identified within 30 days of the index endovascular procedure, combined with requiring dialysis for > 4 weeks
Renal function deterioration | Time of Surgery through Year 10
  New onset of a decrease in eGFR > 30% following treatment when compared to baseline eGFR.
Device integrity events | Time of Surgery through Year 10
  wire fractures, stent kinking, disruption/tears in the graft component, or stent compression or invagination identified through imaging analysis
Reintervention | Time of Surgery through Year 10
  Additional surgical or interventional procedure related to the treated disease / index lesion, the registry device, or to the treatment / procedure.

SECONDARY OUTCOMES:
Characterization of remote data collection to supplement follow-up activities | Time of Surgery through Year 10
  An exploratory description intended to assign significance to an increasingly used method of participant engagement to assess utilization, frequency by time, outcomes, contribution to total follow-up, need for elevation of care
New onset buttock claudication / erectile dysfunction | Time of Surgery through Year 1
  Patient reported

CONTACTS AND LOCATIONS:
Overall Officials: S. Han, Principal Investigator — University of Southern California
Locations (74):
- United States (45):
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - University of California - Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California
  - Mount Sinai Vascular Institute, Miami Beach, Florida
  - University of South Florida, Tampa, Florida
  - VA Medical Center- Atlanta, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - McLaren Heatlh Care Corporation, Bay City, Michigan
  - Corewell Health Medical Group West, Grand Rapids, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Cox Health, Springfield, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University at Buffalo, Research Foundation, Buffalo, New York
  - Mission Hospital, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Universtiy Medical Center, Durham, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist, Winston-Salem, North Carolina
  - University Hospitals - Cleveland Medical Center, Cleveland, Ohio
  - Portland VA Health Care System, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health-Upstate, Greenville, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - HCA Healthcare Research Institute/Columbia Medical Center of Plano, Plano, Texas
  - Baylor Scott and White, Plano, Texas
  - Intermountain Health, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Inova Health Care Services, Falls Church, Virginia
  - Sentara Heart Hospital, Norfolk, Virginia
  - CAMC Health and Education and Research Institute, Inc, Charleston, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Gold Coast Hospital and Health Services, Southport, Queensland
  - Flinders Medical Centre (Vascular Unit), Bedford Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth
  - Royal Prince Alfred Hospital, Sydney
- Medizinische Universitat Wien, Vienna, Austria
- Finland (3):
  - Helsinki University Hospital (HYKS III), Helsinki
  - Wellbeing Services County of Pirkanmaa Tampere University Hospital, Tampere
  - Wellbeing Services County of Pirkanmaa, Tampere
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (5):
  - Azienda Ospedaliero Universitaria delle Marche Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero Universitaria Policlinico di Bari, Bari
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AOU Città della Salute e della Scienza di Torino Ospedale S.Giovanni Battista- Molinette, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Netherlands (3):
  - Amsterdam UMC Research BV, Amsterdam
  - Stichting Elisabeth-Tweesteden Ziekenhuis, Tilburg
  - VieCuri Medical Center, Venlo
- New Zealand (2):
  - Clinical Trials New Zealand Limited - Waikato Hospital, Hamilton, Waikato Region
  - Auckland District Health Board Charitable Trust, Auckland
- Uniwersytecki Szpital Kliniczny NR 1 W Lublinie, Lublin, Poland
- Spain (2):
  - Hospital De La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (4):
  - University Hospitals of Leicester NHS Trust, Leicester
  - Countess of Chester Hospital NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust, St. Mary's Hospital, London
  - St Thomas Hospital - Guys and St. Thomas' NHS, London

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared will be pseudo-anonymized with subject names and birthdates removed, but information such as procedure date will not.
Time Frame: Sharing of IPD will not routinely be performed and is contingent on an assessment of the researcher's proposal for novelty or value in advancing educational, quality or medical practice objectives in use of this data.
Access Criteria: See above